CLINICAL TRIAL: NCT01561755
Title: A Double-Blind, Placebo Controlled Study of Intravenous Immunoglobulin for HIV-Associated Myelopathy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: David M. Simpson (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor-Investigator, David M. Simpson, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 10-1108; HS#: 11-02029
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: HIV-associated Myelopathy
Keywords: HIV associated myelopathy
MeSH Terms: interventions — Immunoglobulins, Intravenous; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous Immunoglobulin (Experimental): Intravenous Immunoglobulin - 2gr/kg over 2 days of Privigen®
  Interventions: Drug: Intravenous Immunoglobulin
- Placebo (Placebo Comparator): Saline 2gr/kg over 2 days of saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous Immunoglobulin — Intravenous Immunoglobulin - 2gr/kg over 2 days of Privigen®
  Other Names: Privigen®; IVIG
  Arms: Intravenous Immunoglobulin
Drug: Placebo — Placebo - 2gr/kg over 2 days of saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Intravenous Immunoglobulin (IVIG) is an effective treatment for HIV associated myelopathy.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether or not intravenous immunoglobulin (lVlg), brand name Privigen, is effective in treating a disorder called HIV-associated myelopathy (HIVM). This drug is currently not approved by the Food and Drug Administration (FDA) for treating this disorder.

HIVM is a spinal cord disease that occurs at any stage of HIV infection. It is not known what causes this condition, but symptoms can include weakness in the lower body and problems with frequent urination or problems with bowel function, trouble walking or performing sexually.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of HIV infection.
* Age ≥ 18
* Males and females are eligible. Subjects must agree to practice birth control or abstinence. Females of child-bearing potential must have a negative urine pregnancy within 14 days prior to study entry.
* Adequate baseline organ function including the following laboratory values within 14 days prior to study entry:
* Adequate liver function with ALT, AST and alkaline phosphatase ≤ 5 times upper limit of normal (ULN).
* Total bilirubin ≤ 2.5 mg/dL Creatinine < 2.3 Serum vitamin B12 level ≥ 200 pg/ml
* Diagnosis of HIVM by a neurologist - defined as:
* - Presence of at least two of the following symptoms:
* - Paresthesias and/or numbness in the lower extremities or in all four limbs; Weakness of the limbs, with predominance in the lower extremities; Unsteady, stiff or uncoordinated gait; Sensation of electrical shock through the back or the legs upon flexion of the neck (L'Hermitte's sign); Stiffness or spasm in the lower extremities; Urinary frequency, urgency, incontinence or retention; Fecal incontinence or retention; Sexual dysfunction with erectile impairment in men;
* - Presence of at least two of the following neurologic signs:
* - Reduction in vibratory or position sensation in the lower extremities; Hyperactive deep tendon reflexes; Abnormal response to plantar stimulation (Babinski sign); Presence of L'Hermitte sign (electrical-type sensation down the back, provoked by flexion of the neck); Weakness in the lower extremities or in all four limbs; Spastic or ataxic gait
* Antiretroviral regimen stable 2 months prior to the entry of the study.

Exclusion Criteria:

* Presence of acute, active, opportunistic infection, except oral thrush, orogenital or rectal herpes and MAI bacteremia within 2 weeks before randomization.
* Evidence of another contributing cause for myelopathy.
* Women who are pregnant, breast-feeding or planning a pregnancy.
* Active abuse of drugs or alcohol, which in the opinion of the investigator would interfere with the subject's ability to comply with the protocol.
* Any neurologic or systemic conditions, which in the opinion of the investigator would interfere with the evaluation of the subject.
* Presence of significant cardiac, pulmonary or renal disease that would place the subject at risk for the fluid and protein load of IVIg.
* History of hypersensitivity to immunoglobulin, or IgA deficiency; Vaccination with live viruses within the past 90 days; Patients receiving IVIg or other immunomodulatory agent (cyclosphosphamide, azathioprine, corticosteroids, tacrolimus, cyclosporine, OKT3, plasma exchange, alpha, beta or gamma interferon) within the past 3 months.
* Patients in whom muscle dynamometry can not be performed for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Simpson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three main sources: the clinical NeuroAIDS practices of the investigators; pre-existing observational research studies (Manhattan HIV Brain Bank and the CNS HIV Antiretroviral Effects Research (CHARTER)); and via a referral network of regional HIV care providers. for a total of four years 2012-2016.
Period: Overall Study
Arm/Group | Intravenous Immunoglobulin | Placebo
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Immunoglobulin | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 48 [29 to 69] | 58 [29 to 68] | 48 [29 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Number of participant with undetectable Viral Load [Count of Participants; unit: Participants] — Number of participants with undetectable viral load <20 copies/ml
  Participants | 1 | 0 | 1
mean CD4+ [Mean (Standard Deviation); unit: cells/mm^3] | 620 (223) | 564 (270) | 592 (212)

OUTCOME MEASURES:

1. Primary Outcome: Strength Scores
Description: Strength score as measured by pounds of force sustained in lower extremity strength.
Time Frame: at 2 months
Measure: Mean (Standard Deviation); unit: pounds of force
Arm/Group | Intravenous Immunoglobulin | Placebo
Number analyzed (Participants) | 6 | 5
pounds of force
  Hip Flexion | 14.0 (32.7) | 1.9 (13.4)
  Knee Flexion | 12.4 (14.4) | 10.3 (14.5)
  Ankle Dorsiflexion | 1.7 (8.2) | -6.0 (5.2)
  Lower extremity - sum of all three | 28.2 (49.2) | 6.2 (28.9)

2. Secondary Outcome: Walking Test
Description: 2 minute walking test
Time Frame: at 2 months
Population: One participant in placebo group in wheelchair and unable to complete the walking test
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Intravenous Immunoglobulin | Placebo
Number analyzed (Participants) | 6 | 4
meters | 93.49 (42.57) | 112.08 (102.00)

3. Secondary Outcome: Urinary Function
Description: 0 = Normal bladder function, 1 = Asymptomatic on current treatment, 2 = Urinary frequency, hesitancy, urgency, with no incontinence, 3 = Occasional urinary incontinence (once or more during the last month but not every week) or intermittent catheterization, 4 = Frequent urinary incontinence, or occasional incontinence despite regular catheterization, 5 = Daily urinary incontinence or permanent catheter
Time Frame: 2 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intravenous Immunoglobulin | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | 2.6 [0 to 5] | 2.5 [0 to 5]

4. Secondary Outcome: Bowel Function
Description: 0 = No bowel problems, 1 = Asymptomatic on current drug tx or constipation not requiring any tx, 2 = Constipation requiring laxative or suppositories or fecal urgency, 3 = Constipation requiring the use of an enema, 4 = Constipation requiring manual evacuation of stools or occasional fecal incontinence (once or more during the last month but not every week, 5 = Weekly fecal incontinence
Time Frame: 2 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intravenous Immunoglobulin | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | 1.3 [0 to 5] | 2.07 [0 to 5]

5. Secondary Outcome: Hughes Function Score
Description: 0 = Normal strength; 1 = minor symptoms but capable of running; 2 = The subject is able to walk 30 ft. but unable to run; 3 = The subject is able to walk 30 ft. with the assistance of one person; 4 = A walker or cane; 5 = The subject is unable to walk.
Time Frame: at 2 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intravenous Immunoglobulin | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | 3 [2 to 4] | 3.2 [1 to 5]

6. Secondary Outcome: Impression of Change Score - Participant
Description: The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment 1. Marked improvement; 2 Moderate Improvement; 3 Minimal Improvement; 4 No Change; 5 Minimal Worsening; 6 Moderate Worsening; 7 Marked worsening
Time Frame: at 2 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intravenous Immunoglobulin | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | 3.58 [2 to 5] | 3.7 [2 to 4]

7. Secondary Outcome: Impression of Change Score - Clinician
Description: The clinician measure of Global Impression of Change reflects the clinician's view about the efficacy of treatment as measured by 1. Marked improvement; 2 Moderate Improvement; 3 Minimal Improvement; 4 No Change; 5 Minimal Worsening; 6 Moderate Worsening; 7 Marked worsening
Time Frame: at 2 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intravenous Immunoglobulin | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | 3.58 [2 to 5] | 4 [3 to 5]

ADVERSE EVENTS:
Arm/Group | Intravenous Immunoglobulin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Immunoglobulin (N=6) | Placebo (N=6)
Mild headache (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment difficult with the widespread availability of IVIG which can be prescribed in an "off-label" fashion, the low incidence of new HIVM cases and a reluctance of this patient population to undergo randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes